CLINICAL TRIAL: NCT04670679
Title: An Open-Label, Multi-Center Phase 1/1b Dose Escalation and Expansion Study of ERAS-601 SHP2 Inhibitor as a Monotherapy and in Combination With Other Anti-Cancer Therapies in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Dose Escalation/Expansion Study of ERAS-601 in Patients With Advanced or Metastatic Solid Tumors
Acronym: FLAGSHP-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Erasca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-601-01
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: SHP2; PTPN11; solid tumor; advanced solid tumor; metastatic solid tumor; neoplasms; solid malignancies; targeted therapy; colorectal cancer; CRC; head and neck squamous cell carcinoma; HPV Negative HNSCC; molecular alterations; cetuximab; Erbitux; Chordoma
MeSH Terms: conditions — Noonan Syndrome; Neoplasm Metastasis; Neoplasms; Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Chordoma | interventions — Cetuximab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation (Part A): ERAS-601 monotherapy (Experimental): ERAS-601 monotherapy will be administered in sequential ascending doses to study participants with advanced or metastatic solid tumors until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-601
- Dose Escalation (Part B): ERAS-601 monotherapy (Experimental): ERAS-601 monotherapy will be administered in sequential ascending doses to study participants with advanced or metastatic solid tumors until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-601
- Dose Escalation (Part C): ERAS-601 monotherapy (Experimental): ERAS-601 will be administered in sequential ascending doses to study participants with advanced or metastatic solid tumors until unacceptable toxicity, disease progression or withdrawal of consent.
  Interventions: Drug: ERAS-601
- Dose Escalation and Dose Expansion (Part D): ERAS-601 in combination with cetuximab (Experimental): ERAS-601 will be administered in sequential ascending doses with cetuximab to study participants with advanced metastatic solid tumors until unacceptable toxicity, disease progression or withdrawal of consent. Once the combination therapy recommended dose has been determined, this will be administered to study participants with HPV negative advanced or metastatic head and neck squamous cell carcinoma (HNSCC) or colorectal cancer (CRC).
  Interventions: Drug: ERAS-601; Drug: Cetuximab
- Dose Escalation and Dose Expansion (Part E): ERAS-601 in combination with pembrolizumab (Experimental): ERAS-601 will be administered in sequential ascending doses with pembrolizumab to study participants with advanced metastatic solid tumors until unacceptable toxicity, disease progression or withdrawal of consent. Once the combination therapy recommended dose has been determined, this will be administered to study participants with HPV negative advanced or metastatic head and neck squamous cell carcinoma (HNSCC) or non small cell lung cancer (NSCLC).
  Interventions: Drug: ERAS-601; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ERAS-601 — Administered orally
Drug: Cetuximab — Administered via intravenous infusion
  Other Names: Erbitux
  Arms: Dose Escalation and Dose Expansion (Part D): ERAS-601 in combination with cetuximab
Drug: Pembrolizumab — Administered via intravenous infusion
  Other Names: Keytruda
  Arms: Dose Escalation and Dose Expansion (Part E): ERAS-601 in combination with pembrolizumab

SUMMARY:
* To evaluate the safety and tolerability of escalating doses of ERAS-601 when administered as a monotherapy and in combination with other cancer therapies in study participants with advanced or metastatic solid tumors.
* To determine the Maximum Tolerated Dose (MTD) and/or recommended dose (RD) of ERAS-601 when administered as a monotherapy and in combination with other cancer therapies.
* To characterize the pharmacokinetic (PK) profile of ERAS-601 when administered as a monotherapy and in combination with other cancer therapies.
* To evaluate the antitumor activity of ERAS-601 when administered as a monotherapy and in combination with other cancer therapies.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1/1b, open-label, multicenter clinical study of ERAS-601 as a monotherapy and in combination with other cancer therapies. The study will commence with dose escalation of ERAS-601 monotherapy, followed by dose escalation of ERAS-601 in combination with other cancer therapies. Once the monotherapy MTD and/or RD has been determined, then dose expansion of ERAS-601 monotherapy may commence with enrollment of study participants with advanced or metastatic solid tumors harboring specific molecular alterations. Once the combination therapy MTD and/or RD has been determined, then dose expansion of that combination may commence with enrollment of study participants with advanced or metastatic solid tumors harboring specific molecular alterations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing and able to give written informed consent
* Have histologically or cytologically confirmed advanced or metastatic solid tumor
* There is no available standard systemic therapy available for the patient's tumor histology and/or molecular biomarker profile; or standard therapy is intolerable, not effective, or not accessible; or patient has refused standard therapy
* Able to swallow oral medication
* Have Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* Adequate cardiovascular, hematological, liver, and renal function
* Willing to comply with all protocol-required visits, assessments, and procedures

Exclusion Criteria:

* Previous treatment with a SHP2 inhibitor
* Documented PTPN11 mutations
* Is currently receiving another study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of the first dose of ERAS-601
* Received prior palliative radiation within 7 days of Cycle 1, Day 1
* Have primary central nervous system (CNS) disease or known active CNS metastases and/or carcinomatous meningitis
* Prior surgery (e.g., gastric bypass surgery, gastrectomy) or gastrointestinal dysfunction (e.g., Crohn's disease, ulcerative colitis, short gut syndrome) that may affect drug absorption
* Active, clinically significant interstitial lung disease or pneumonitis
* History of thromboembolic or cerebrovascular events ≤ 12 weeks prior to the first dose of study treatment
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO
* Have any underlying medical condition, psychiatric condition, or social situation that, in the opinion of the Investigator, would compromise study administration as per protocol or compromise the assessment of AEs
* Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Study Day 1 up to Day 29
  Based on toxicities observed
Maximum tolerated dose (MTD) | Study Day 1 up to Day 29
  Based on toxicities observed
Recommended dose (RD) | Study Day 1 up to Day 29
  Based on toxicities observed
Adverse Events | Assessed up to 24 months from time of first dose
  Incidence and severity of treatment-emergent AEs and serious AEs
Plasma concentration (Cmax) | Study Day 1 up to Day 29
  Maximum plasma concentration of ERAS-601 and cetuximab or pembrolizumab (if applicable)
Time to achieve Cmax (Tmax) | Study Day 1 up to Day 29
  Time to achieve maximum plasma concentration of ERAS-601 and cetuximab or pembrolizumab (if applicable)
Area under the curve | Study Day 1 up to Day 29
  Area under the plasma concentration-time curve of ERAS-601 and cetuximab or pembrolizumab (if applicable)
Half-life | Study Day 1 up to Day 29
  Half-life of ERAS-601 and cetuximab or pembrolizumab (if applicable)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Duration of Response (DOR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Time to Response (TTR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1

OTHER OUTCOMES:
Pharmacodynamic assessment | Assessed up to 24 months from time of first dose
  Assessment of phosphorylated ERK (pERK) inhibition in PBMCs or tumor tissue by IHC or immunofluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: Les Brail, PhD, Study Director — Clinical Development
Locations (14):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sarah Cannon Research Institute (Florida Cancer Specialists), Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute (Tennessee Oncology), Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No